CLINICAL TRIAL: NCT01217008
Title: A Phase 1 Safety Study of GRNOPC1 in Patients With Neurologically Complete, Subacute, Spinal Cord Injury
Brief Title: Safety Study of GRNOPC1 in Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lineage Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP35A007
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2014-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; GRNOPC1
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRNOPC1 (Experimental): Subjects who receive an injection of GRNOPC1
  Interventions: Biological: GRNOPC1

INTERVENTIONS:
Biological: GRNOPC1 — One injection of 2 million GRNOPC1 cells.

SUMMARY:
The purpose of the study is to evaluate the safety of GRNOPC1 administered at a single time-point between 7 and 14 days post injury, inclusive, to patients with neurologically complete spinal cord injuries (SCI).

ELIGIBILITY:
Major Inclusion Criteria:

* Neurologically complete, traumatic SCI (ASIA Impairment Scale A), zone of partial preservation < 5 levels
* Last fully preserved neurological level from T-3 through T-11
* From 18 through 65 years of age at time of injury
* Single spinal cord lesion
* Informed consent for this protocol and the companion long term follow-up protocol must be provided and documented (i.e., signed informed consent forms) no later than 11 days following injury
* Able to participate in an elective surgical procedure to inject GRNOPC1 7-14 days following SCI

Major Exclusion Criteria:

* SCI due to penetrating trauma
* Traumatic anatomical transection or laceration of the spinal cord
* Any concomitant injury or pre-existing condition that interferes with the performance, interpretation or validity of neurological examinations
* Inability to communicate effectively with neurological examiner
* Significant organ damage or systemic disease that would create an unacceptable risk for surgery or immunosuppression
* History of any malignancy
* Pregnant or nursing women
* Body mass index (BMI) > 35 or weight > 300 lbs.
* Active participation in another experimental procedure/intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety | One year
  The primary endpoint is safety, as measured by the frequency and severity of adverse events within 1 year (365 days) of GRNOPC1 injection that are related to GRNOPC1, the injection procedure used to administer GRNOPC1, and/or the concomitant immunosuppression administered.

SECONDARY OUTCOMES:
Neurological function | One year
  The secondary endpoint is neurological function as measured by sensory scores and lower extremity motor scores on International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) examinations.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University/Santa Clara Valley Medical Center, Palo Alto/San Jose, California
  - Shepherd Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Maryland Medical Center/Kernan Orthopaedics and Rehabilitation Hospital, Baltimore, Maryland
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The Medical College of Wisconsin, Milwaukee, Wisconsin